CLINICAL TRIAL: NCT02395029
Title: Evaluate the Safety and Feasibility of Injecting Placental Matrix-Derived Mesenchymal Stem Cells Into the Penis to Treat the Symptoms of Peyronie's Disease
Brief Title: Evaluate the Safety and Feasibility of Injecting PMD-MSC Into the Penis to Treat the Symptoms of PD
Acronym: PMD-MSC-PD-01
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Melissa Marchand (Other)
Responsible Party: Sponsor-Investigator, Melissa Marchand, PA-C, Z Urology
Organization: Z Urology (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PMD-MSC-PD-01
Record Dates: First submitted 2015-03-09; First posted 2015-03-20 (Estimated); Last update posted 2015-03-20 (Estimated); Status verified 2015-03

CONDITIONS: Peyronie's Disease
Keywords: PD
MeSH Terms: conditions — Penile Induration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Injection of PMD-MSCs into the penis (Experimental): Subjects will receive an initial injection of 1.0cc of Placental Matrix-Derived Mesenchymal Stem Cells (PMD-MSCs). Subjects will be eligible for re-injection at 3 months and/or 6 months as determined by the clinician based on ultrasound guided measurements of penile plaque(s) post treatment and on patient reported treatment satisfaction.
  Interventions: Biological: Placental Matrix-Derived Mesenchymal Stem Cells (PMD-MSCs)

INTERVENTIONS:
Biological: Placental Matrix-Derived Mesenchymal Stem Cells (PMD-MSCs)
  Other Names: Ovation

SUMMARY:
Prospective, open labeled, non-randomized, study to be conducted at a single center. Ten subjects will undergo an injection of Placental Matrix-Derived Mesenchymal Stem Cells (PMD-MSCs) into the penis for the treatment of Peyronie's Disease. Follow up visits will be conducted at 6 weeks, 3 months, 6 months, and 12 months. Subjects will be eligible for re-injection at 3 months and/or 6 months as determined by the clinician based on patient reported treatment satisfaction.

DETAILED DESCRIPTION:
Symptoms of Peyronie's disease include penile pain and curvature of the penis that prevents penetration and/or causes erectile dysfunction (ED). It is characterized by plaques that form along the top or bottom side of the penis inside the tunica albuginea; the plaque begins as a localized inflammation then develops into a hardened scar. Cases can range from mild to severe. In several cases, the hardened plaque reduces flexibility, causing the penis to curve during erection. The sexual problems as a result can lower a man's self-esteem and interfere with a couple's physical and emotional relationship.

The cause is unknown; however, possibilities include trauma, inherited conditions, Vitamin E deficiency, diabetes, and vascular disease.

Conservative treatments used in the acute phase (initial onset of symptoms) include oral therapies. Vitamin E and antioxidants can decrease the build-up of harmful chemicals that can cause injury to tissue. It is often used as the traditional treatment; it is inexpensive and with proper dosing, there are minimal side effects. Other oral agents include Potaba (aminobenzoates potassium); however, it is expensive ($1000 per year) and has associated gastrointestinal side effects.

Other therapies involve injections directly in the plaques (intralesional) with chemicals such as collagenase or calcium-channel blockers.

Surgical therapies are offered once the disease is stable (symptoms present for one year). Invasive surgical options consist of correction of the penile curvature or the placement of a penile prosthesis to straighten the penis to allow for erections.

Mesenchymal stem cells (MSCs) have been used for a variety of medical treatments to repair and regenerate acute and chronically damaged tissues. These cells have the potential to repair human tissue by forming cells of mesenchymal origin, such as cartilage, bone, fat, muscle, and blood vessels. Most research has focused on bone marrow derived stem cells (BMC) however the process for harvesting the cells is invasive, painful, and yields a low cell count. The human placenta offers an alternative source form MSCs. Placental Matrix-Derived Mesenchymal Stem Cells (PMD-MSCs) are compromised of a novel cellular repair matrix derived from placental mesenchyme. Mesenchyme is the meshwork of embryonic connective tissue in the mesoderm, from which are formed the muscular and connective tissues of the body and also the blood vessels. PMD-MSCs provide the extracellular matrix viable mesenchymal stem cells (MSCs) that coordinate the tissue repair process, regenerative growth factors, and anti-inflammatory cytokines required to regenerate the damaged vasculature of the penile corpora.

The research proposed here will establish the safety and feasibility of utilizing intracavernosal, intralesional injections of PMD-MSCs to treat Peyronie's disease with the intent of avoiding surgery.

ELIGIBILITY:
Inclusion Criteria:

1. acquired penile curvature >15 and <90 degrees associated with palpable penile plaque on physical examination
2. 1 or 2 penile plaque at screening

Exclusion Criteria:

1. taking the medication Coumadin
2. unable to achieve adequate erection with penile injection to access degree of curvature
3. undergone definitive treatment for prostate cancer, bladder cancer, or other pelvic malignancies including surgery, external beam radiation therapy, brachytherapy, cryotherapy
4. prior history of prostate cancer, hematologic disorders, chronic liver disease including cirrhosis and hepatitis C, disorders affecting the immune system, including infection with the human immunodeficiency virus, or psychiatric disorder including major depression, schizophrenia, bipolar disease
5. history of cerebrovascular accident, history of deep venous thrombosis within the past 5 years or history of untreated or severe sleep apnea
6. clinically significant abnormal lab results that would put the subject at increased risk or compromise the integrity of the study data, in the opinion of the investigator
7. received any other investigational drug within 30 days

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2013-08; Primary Completion 2014-12 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Peak Systolic Velocity without trimix (cm/s) | Baseline
Peak Systolic Velocity without trimix (cm/s) | 6 weeks
Peak Systolic Velocity without trimix (cm/s) | 3 months
Peak Systolic Velocity without trimix (cm/s) | 6 months
Peak Systolic Velocity without trimix (cm/s) | 12 months

SECONDARY OUTCOMES:
End Diastolic Velocity without trimix (cm/s) | Baseline
End Diastolic Velocity without trimix (cm/s) | 6 weeks
End Diastolic Velocity without trimix (cm/s) | 3 months
End Diastolic Velocity without trimix (cm/s) | 6 months
End Diastolic Velocity without trimix (cm/s) | 12 months

OTHER OUTCOMES:
Peak Systolic Velocity with trimix (cm/s) | Baseline
Peak Systolic Velocity with trimix (cm/s) | 6 weeks
Peak Systolic Velocity with trimix (cm/s) | 3 months
Peak Systolic Velocity with trimix (cm/s) | 6 months
Peak Systolic Velocity with trimix (cm/s) | 12 months
End Diastolic Velocity with trimix (cm/s) | Baseline
End Diastolic Velocity with trimix (cm/s) | 6 weeks
End Diastolic Velocity with trimix (cm/s) | 3 months
End Diastolic Velocity with trimix (cm/s) | 6 months
End Diastolic Velocity with trimix (cm/s) | 12 months
Rigidity test (Pass or Fail) | Baseline
Rigidity test (Pass or Fail) | 6 weeks
Rigidity test (Pass or Fail) | 3 months
Rigidity test (Pass or Fail) | 6 months
Rigidity test (Pass or Fail) | 12 months
Stretched Penile Length before trimix (cm/s) | Baseline
Stretched Penile Length before trimix (cm/s) | 6 weeks
Stretched Penile Length before trimix (cm/s) | 3 months
Stretched Penile Length before trimix (cm/s) | 6 months
Stretched Penile Length before trimix (cm/s) | 12 months
Post Penile Width with trimix | Baseline
Post Penile Width with trimix | 6 weeks
Post Penile Width with trimix | 3 months
Post Penile Width with trimix | 6 months
Post Penile Width with trimix | 12 months
International Index of Erectile Function (IIEF) | Baseline
International Index of Erectile Function (IIEF) | 6 weeks
International Index of Erectile Function (IIEF) | 3 months
International Index of Erectile Function (IIEF) | 6 months
International Index of Erectile Function (IIEF) | 12 months
#1 Penile Plaque (Location) Size (mm^3) | Baseline
#1 Penile Plaque (Location) Size (mm^3) | 6 weeks
#1 Penile Plaque (Location) Size (mm^3) | 3 months
#1 Penile Plaque (Location) Size (mm^3) | 6 months
#1 Penile Plaque (Location) Size (mm^3) | 12 months
#2 Penile Plaque (Location) Size (mm^3) | Baseline
#2 Penile Plaque (Location) Size (mm^3) | 6 weeks
#2 Penile Plaque (Location) Size (mm^3) | 3 months
#2 Penile Plaque (Location) Size (mm^3) | 6 months
#2 Penile Plaque (Location) Size (mm^3) | 12 months
#3 Penile Plaque (Location)Size (mm^3) | Baseline
#3 Penile Plaque (Location)Size (mm^3) | 6 weeks
#3 Penile Plaque (Location)Size (mm^3) | 3 months
#3 Penile Plaque (Location)Size (mm^3) | 6 months
#3 Penile Plaque (Location)Size (mm^3) | 12 months
Penile Curvature Angle (degrees) | Baseline
Penile Curvature Angle (degrees) | 6 weeks
Penile Curvature Angle (degrees) | 3 months
Penile Curvature Angle (degrees) | 6 months
Penile Curvature Angle (degrees) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael P. Zahalsky, M.D., Principal Investigator — Z Urology
Locations (1):
- Z Urology, Coral Springs, Florida, United States

REFERENCES:
- [Derived] Levy JA, Marchand M, Iorio L, Zribi G, Zahalsky MP. Effects of Stem Cell Treatment in Human Patients With Peyronie Disease. J Am Osteopath Assoc. 2015 Oct;115(10):e8-13. doi: 10.7556/jaoa.2015.124. PMID 26414724